CLINICAL TRIAL: NCT00034645
Title: Prophylaxis Trial in High Risk Allogenic Stem Cell Transplant Recipients With Graft vs. Host Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: C98316; C/I98-316 (Other: Sponsor)
Record Dates: First submitted 2002-05-01; First posted 2002-05-02 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Mycoses
Keywords: Allogenic Stem cell transplantation; Fungal infections
MeSH Terms: conditions — Mycoses

INTERVENTIONS:
Drug: Posaconazole oral suspension

SUMMARY:
This trial is in high risk patients to determine the safety, tolerance and efficacy of posaconazole (POZ) vs. fluconazole in the prophylaxis against development of invasive fungal infections (IFI).

DETAILED DESCRIPTION:
This study is designed to determine the safety, tolerance and efficacy of POZ used as prophylaxis of IFI in high-risk subjects with Grade II-IV acute graft vs. host disease (GVHD) or extensive chronic GVHD. The primary objective is to assess the efficacy of SCH56592 vs fluconazole in preventing proven or probable IFI within the time period from randomization to 16 weeks after the start of treatment with study drug.

ELIGIBILITY:
Inclusion Criteria:

* Hematopoietic progenitor cell transplant subjects with chronic or Grade II-IV acute GVHD being treated with high dose immunosuppressive therapy.
* One of the following to the subject's prior immunosuppressive regimen:

  1. at least 1mg per kg per day of methylprednisolone or equivalent,
  2. Antithymocyte globulin (ATG) for the therapy of acute GVHD,
  3. Tacrolimus, mycophenolate mofetil, or other steroid-sparing immunosuppressive regimen.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 1999-01; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

REFERENCES:
- [Derived] Ullmann AJ, Lipton JH, Vesole DH, Chandrasekar P, Langston A, Tarantolo SR, Greinix H, Morais de Azevedo W, Reddy V, Boparai N, Pedicone L, Patino H, Durrant S. Posaconazole or fluconazole for prophylaxis in severe graft-versus-host disease. N Engl J Med. 2007 Jan 25;356(4):335-47. doi: 10.1056/NEJMoa061098. PMID 17251530
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html